CLINICAL TRIAL: NCT05801185
Title: Single Nuclei Sequencing in Human Skeletal Muscle After Unloading
Acronym: ULLS23
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Rodrigo Fernandez Gonzalo, PhD and docent (Associate Professor), Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Dnr 2022-04662-01
Record Dates: First submitted 2023-03-13; First posted 2023-04-06 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Unilateral Lower Limb Suspension
Keywords: ULLS; single nuclei RNA sequencing; Skeletal muscle

STUDY DESIGN:
Intervention Model Description: Participants will perform a 5-day unloading intervention using the ULLS model. Short-length crutches, aided by handgrip and forearm support distal to the elbow will be used to assist in any upright or ambulatory activity. One foot (randomized in a counterbalance manner) will be equipped with a shoe having a 10-cm thick sole, which permits the unloaded limb to move passively about the hip joint while adopting a near straight position.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unilateral lower limb suspension (Experimental): Participants will perform a 5-day unloading intervention using the ULLS model. Short-length crutches, aided by handgrip and forearm support distal to the elbow will be used to assist in any upright or ambulatory activity. One foot (randomized in a counterbalance manner) will be equipped with a shoe having a 10-cm thick sole, which permits the unloaded limb to move passively about the hip joint while adopting a near straight position.
  Interventions: Other: Unilateral lower limb suspension

INTERVENTIONS:
Other: Unilateral lower limb suspension — Participants will perform a 5-day unloading intervention using the ULLS model. Short-length crutches, aided by handgrip and forearm support distal to the elbow will be used to assist in any upright or ambulatory activity. One foot (randomized in a counterbalance manner) will be equipped with a shoe having a 10-cm thick sole, which permits the unloaded limb to move passively about the hip joint while adopting a near straight position.

SUMMARY:
Injuries often require people to undergo some degree of limb immobilization. This comes at a high cost in terms of muscle mass and function losses. At the molecular level, it is completely unknown how the different cells in the muscle respond to this complete lack of mechanical stimuli.

The investigators will explore cell type specific changes in skeletal muscle after a short period of unloading, and specifically examine the behavior of myogenic stem cells with particular attention to potential unloading-induced maturation into fast- or slow-twitch muscle fibers.

Ten healthy young participants will perform a 5-day Unilateral Lower Limb Suspension (ULLS) intervention, where one leg is continuously subjected to unloading, i.e., lack of mechanical stimuli. Before and after the ULLS period, participants will perform muscle function testing and MRI scans to assess muscle size in the lower limbs. Immediately after the ULLS, two muscle biopsies will be obtained, one from each leg. The tissue will be employed for single-nuclei RNA sequencing analysis and immunohistochemistry experiments.

This project will be the first to analyze cell type specific changes induced by complete, short-term lack of mechanical stimuli in skeletal muscle. This will add a new dimension to the understanding of the processes directing this type of muscle atrophy (i.e., muscle loss in otherwise healthy individuals) and thus help to develop effective countermeasures to offset muscle changes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adult men

Exclusion Criteria:

* An age younger than 18 or older than 40 years
* Contraindications to magnetic resonance imaging (MRI)
* Contraindications to maximal intensity resistance exercise
* Contraindications to unloading (i.e., ULLS)
* Very high physical activity levels (determined using a standard Godin Leisure-Time Exercise Questionnaire (GLTEQ))
* Hypertension (>140/90 mm Hg)
* History of malignancy
* History of coagulation dysfunction
* History of musculoskeletal or neurological disorders
* History of cardiovascular disease
* History of cerebrovascular disease
* History of respiratory disease
* History of gastrointestinal disease
* History of renal disease
* History of past or present condition requiring long-term drug prescriptions.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Single nuclei RNA sequencing | Immediately after the 5-day unilateral unloading intervention
  Single nuclei RNA sequencing from skeletal muscle (m. vastus lateralis) from both legs

SECONDARY OUTCOMES:
Muscle mass | Before and immediately after the 5-day unloading intervention
  Muscle volume of quadriceps muscle group (and individual muscles) assessed by MRI in both legs
Concentric isokinetic torque of knee extensor muscles | Before and immediately after the 5-day unloading intervention
  Concentric isokinetic torque of knee extensor muscles at 30°/s, 90°/s, 180°/s and 300°/s, measured with an isokinetic dynamometer unilaterally in both legs
Isometric torque of knee extensor muscles | Before and immediately after the 5-day unloading intervention
  Isometric torque of knee extensor muscles at 60° knee flexion, measured with an isokinetic dynamometer unilaterally in both legs

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No